CLINICAL TRIAL: NCT03400631
Title: Changes in Cytokines After Masked Intraarticular Injection of Dextrose or Aspiration Only in Stage IV Knee Osteoarthritis
Brief Title: Changes in Cytokine Levels After Dextrose Injection in Stage IV Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisiatria y Traumatología (Other)
Collaborators: American Association of Orthopaedic Medicine (Unknown)
Responsible Party: Principal Investigator, Gaston Andres Topol, Gaston Topol, M.D., Principal Investigator, Fisiatria y Traumatología
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AAFOYT
Record Dates: First submitted 2017-10-25; First posted 2018-01-17 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Cytokine
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The first two weeks of this study involve two groups with a crossover at 1 week. From two weeks on, there is a single arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only of above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose 0. Aspiration 1 week. (Experimental): Dextrose injection given at time 0, at 1 week aspiration only, and then open label injection of dextrose at 0, 1, 2, 3, 4, 5, and 6 months.
  Interventions: Drug: Dextrose 0; Drug: Aspiration 1
- Aspiration 0. Dextrose 1 week. (Experimental): Aspiration only at time 0. Dextrose injection given at 1 week, and then open label injection of dextrose at 0, 1, 2, 3, 4, 5, and 6 months.
  Interventions: Drug: Aspiration 0; Drug: Dextrose 1

INTERVENTIONS:
Drug: Dextrose 0 — Dextrose injection at time 0
  Arms: Dextrose 0. Aspiration 1 week.
Drug: Aspiration 0 — Aspiration only at time 0
  Arms: Aspiration 0. Dextrose 1 week.
Drug: Dextrose 1 — Dextrose injection at week 1
  Arms: Aspiration 0. Dextrose 1 week.
Drug: Aspiration 1 — Aspiration only at week 1
  Arms: Dextrose 0. Aspiration 1 week.

SUMMARY:
Twenty participants with severe arthritis will be enrolled. For the first week participants will either be injected with dextrose or just have fluid withdrawn for testing. The remaining participants will be given dextrose injection at the end of the week. After one week dextrose injections will be given at one, two, three, four, five, and six months. Fluid will be withdrawn from the knee at time zero, one week, and three months. The hypothesis is that dextrose injection will cause a change in proteins in the knee consistent with improved repair signals, along with improving knee pain and function. .

DETAILED DESCRIPTION:
Participants with stage IV knee osteoarthritis will be evaluated for eligibility and randomized 1 to 1 using an Internet randomization method to ensure random allocation.

At time zero all participants will receive aspiration of their knees from the suprapatellar pouch of 5.5 mL of synovial fluid for cytokine analysis. After that 10 of the participants will receive injection of 10 mL of 12.5% dextrose. The other 10 will receive no injection after aspiration. Pain levels will be measured at time zero, 15 minutes, two hours and 48 hours after aspiration with or without injection to gather information about the time course of analgesia.

At one week all participants will receive aspiration of 2.0 mL from the suprapatellar pouch for cytokine analysis, followed by injection of the remaining 10 participants with dextrose 12.5%. Pain levels will be measured at the same time intervals to complete evaluation of dextrose analgesia.

After two weeks injections will be open label with 10 mills of dextrose 12 and have percent injected at one, two, three, four, five, and six months. At the three month. Another 2 mL of synovial fluid will be sent to the laboratory for cytokine analysis.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain for at least 6 months.
* Clinically diagnosed knee osteoarthritis.
* Weight-bearing radiograph consistent with high-grade medial compartment cartilage loss (Kellgren-Lawrence Grading Scale level IV).
* Confirmation of exposed subchondral bone by high-resolution knee ultrasonography.

Exclusion Criteria:

* Anticoagulation therapy.
* Inflammatory or post-infectious knee arthritis.
* Systemic inflammatory conditions.
* Knee flexion of less than 100 degrees.
* Knee extension of less than 165 degrees.
* Any Valgus
* Varus more than 15 degrees.
* Any knee injection in the past 3 months.
* BMI more than 40
* Gross synovial folds on ultrasound
* Elevation of sed rate, C reactive protein, rheumatoid factor or antinuclear antibody.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Short term change in cytokine levels | Obtained at baseline and 1 week
  Change in cytokine levels from baseline to 1 week
Long term change in cytokine levels | Obtained at baseline and 3 months
  Change in cytokine levels from baseline to 3 months

SECONDARY OUTCOMES:
Post Injection Short Term Pain Course | 0, 15 minutes, 2 hours, and 48 hours after time 0 and 1 week injections
  Numerical rating scale (NRS) 0-10 pain score measured after time 0 and 1 week injections
WOMAC score | Obtained at baseline, 3 and 6 months.
  Western Ontario and McMaster Universities Arthritis Index normalized to 100

CONTACTS AND LOCATIONS:
Overall Officials: Gaston Topol, M.D., Principal Investigator — University of Argentina
Locations (1):
- Gaston Topol, M.D.. Private Office, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
This will be available by request.

REFERENCES:
- [Background] Sit RW, Chung VCh, Reeves KD, Rabago D, Chan KK, Chan DC, Wu X, Ho RS, Wong SY. Hypertonic dextrose injections (prolotherapy) in the treatment of symptomatic knee osteoarthritis: A systematic review and meta-analysis. Sci Rep. 2016 May 5;6:25247. doi: 10.1038/srep25247. PMID 27146849
- [Background] Topol GA, Podesta LA, Reeves KD, Giraldo MM, Johnson LL, Grasso R, Jamin A, Clark T, Rabago D. Chondrogenic Effect of Intra-articular Hypertonic-Dextrose (Prolotherapy) in Severe Knee Osteoarthritis. PM R. 2016 Nov;8(11):1072-1082. doi: 10.1016/j.pmrj.2016.03.008. Epub 2016 Apr 4. PMID 27058744